CLINICAL TRIAL: NCT00656851
Title: Myocardial Function, Free Fatty Acid and Glucose Metabolism in HIV Metabolic Syndrome
Brief Title: Myocardial Function & FFA Metabolism in HIV Metabolic Syndrome
Acronym: WU197
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kevin Yarasheski, Professor of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DK59531 (completed); HRPO 05-0976
Record Dates: First submitted 2008-04-10; First posted 2008-04-11 (Estimated); Results first posted 2013-08-20 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: HIV Infections; Cardiovascular Disease; Insulin Resistance; HIV Lipodystrophy; The Metabolic Syndrome
Keywords: HIV/AIDS; Heart disease; Diabetes; Cardiovascular disease risk; Dyslipidemia; Visceral adiposity; treatment experienced
MeSH Terms: conditions — HIV Infections; Cardiovascular Diseases; Insulin Resistance; Acquired Immunodeficiency Syndrome; Heart Diseases; Diabetes Mellitus; Dyslipidemias | interventions — Pioglitazone; Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone (Active Comparator): Pioglitazone (Actos, 30mg/day for 16 weeks)
  Interventions: Drug: Pioglitazone
- Exercise Training (Active Comparator): Cardiorespiratory and resistance exercise training 3days/wk for 16 weeks
  Interventions: Behavioral: Exercise Training

INTERVENTIONS:
Drug: Pioglitazone — 30mg/day for 16 weeks
  Other Names: Actos
  Arms: Pioglitazone
Behavioral: Exercise Training — Cardiorespiratory and resistance exercise training 3days/wk for 16 weeks
  Other Names: Physical activity; Aerobic exercise; Weight lifting exercise
  Arms: Exercise Training

SUMMARY:
We hypothesize that the hearts of HIV+ people with The Metabolic Syndrome use and oxidize fats and sugars inappropriately, and that this may impair the heart's ability to pump blood. We hypothesize that exercise training or pioglitazone (Actos) will improve fat and sugar metabolism in the hearts of HIV+ people with The Metabolic Syndrome. This study will advance our understanding of cardiovascular disease in HIV+ people, and will test the efficacy of exercise training and pioglitazone for improving insulin resistance, heart metabolism and heart function in this at risk population.

DETAILED DESCRIPTION:
We hypothesize that myocardial free fatty acid and glucose utilization and oxidation rates are dysregulated in HIV+ people with The Metabolic Syndrome in comparison to HIV+ people without The Metabolic Syndrome, and in comparison to HIV-seronegative people with and without The Metabolic Syndrome. We hypothesize that dysregulated myocardial fatty acid and glucose metabolism is associated with impaired heart function (diastolic dysfunction) in HIV+ people with The Metabolic Syndrome. We will use myocardial positron emission tomography, radioactive isotope tracers of palmitate and glucose, and echocardiography to evaluate myocardial metabolism and function. HIV+ people with The Metabolic Syndrome will receive 16wks of exercise training or pioglitazone (Actos), and we will evaluate their potential beneficial effects on myocardial metabolism and function.

ELIGIBILITY:
Inclusion Criteria: All participants both with and without metabolic syndrome:

1. 28-50 years old.
2. Plasma HIV RNA less than 5,000 copies/mL for previous 3 months OR CD4 count greater than 100 cells/µL for previous 3 months.
3. Stable for at least the past 3 months on any HAART regimen.
4. "Normal" blood chemistries for at least 1 month prior to enrollment: platelet count >50,000/mm3, absolute neutrophil count >750/mm3, liver transaminases <2.5x the upper limit of normal (ULN), creatinine <1.3x ULN, albumin >30g/L, creatine kinase <5.9x ULN.

Menstruating women must have a negative urine beta-HCG pregnancy test within 14 days prior to study. To control for potential metabolic effects of alterations in female hormones during the menstrual cycle, all menstruating women will be studied during the follicular phase (serum 17beta-estradiol <165 pg/mL).

Exclusion Criteria:

1. Frank obesity (BMI >35kg/m2).
2. Chronic hepatitis B infection (HB surface antigen positive). Active hepatitis C infection (detectable Hep C RNA). Those who have cleared hepatitis B or C infection are eligible.
3. Diabetes [fasting glucose >125 mg/dL, or fasting insulin >45 µU/mL, or 2-hr glucose >200mg/dL].
4. Medications or agents that regulate glucose metabolism (e.g., insulin-sensitizers, insulin-secretagogues). Lipid lowering agents that regulate lipid metabolism (i.e. fibrate, statin).
5. Gestational diabetes, pregnancy, or nursing mothers.
6. Serum triglycerides ≥ 500 mg/dL.
7. Hypogonadism [total testosterone <200ng/dL (men) or <15ng/dL (women)]; thyroid disorder [TSH <0.2 or >12µIU/mL]; hypercortisolemia [morning cortisol >22µg/dL]. Replacement testosterone or thyroid hormones to normalize abnormal levels is acceptable, as long as treatment and blood levels have been stable for at least 3 months.
8. Use of human growth hormone (hGH) or GH-secretagogues (GH-releasing hormone-peptides) within the previous 3 months.
9. History of serious cardiovascular disease; MI, angina pectoris, heart failure, congenital heart disease, coronary artery disease, coronary artery bypass graft, stroke. Bundle branch block is exclusionary because it limits the interpretability of the resting/exercise ECG. Cardiovascular or physical contraindications to maximal exercise testing on a cycle ergometer.
10. Uncontrolled hypertension (>140/90 mmHg). Certain antihypertensive medications will be permitted (diuretics, ACE inhibitors) as long as the medication, dose, and blood pressure have been stable for at least 3 months.
11. Well-trained athletes (defined as >3 exercise training exposures/week; >30min regimented exercise/exposure maintained for at least the prior 4 weeks).
12. History of or active substance abuse (eg, alcoholism, cocaine, heroin, crack, methamphetamine, phencyclidine).
13. Active secondary infection. Any significant change in chronic suppressive therapy for an opportunistic infection during 1 month prior to enrollment.
14. New serious systemic infection during the 3 weeks prior to enrollment.
15. History of hyperlactatemia or lactic acidosis, esp. with rapid weight loss.
16. Debilitating-painful myopathy or neuropathy that requires 'assistance' to conduct normal activities of daily living (dressing, hygiene, preparing meals, operating a vehicle). These might affect peripheral substrate metabolism.
17. Chronic renal insufficiency/failure or other comorbid conditions (eg. cancer, COPD) that alter metabolism.
18. Pancreatitis, celiac disease, or cirrhosis.
19. Inadequate macronutrient or energy intake, or malabsorptive disorder.
20. Dementia or any condition that would prevent voluntary informed consent or compliance.
21. Other compounds or blinded investigational new drugs that might affect metabolism or confound data interpretation (eg. RU486, interleukin therapy, or cytokine-receptor antagonist).
22. Oral glucocorticoid or corticosteroid use within previous 3 months.

Ages: 28 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2005-09; Primary Completion 2009-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Yarasheski, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Cade WT, Reeds DN, Overton ET, Herrero P, Waggoner AD, Davila-Roman VG, Lassa-Claxton S, Gropler RJ, Soto PF, Krauss MJ, Yarasheski KE, Peterson LR. Effects of human immunodeficiency virus and metabolic complications on myocardial nutrient metabolism, blood flow, and oxygen consumption: a cross-sectional analysis. Cardiovasc Diabetol. 2011 Dec 8;10:111. doi: 10.1186/1475-2840-10-111. PMID 22151886
- [Result] Cade WT, Overton ET, Mondy K, de las Fuentes L, Davila-Roman VG, Waggoner AD, Reeds DN, Lassa-Claxton S, Krauss MJ, Peterson LR, Yarasheski KE. Relationships among HIV infection, metabolic risk factors, and left ventricular structure and function. AIDS Res Hum Retroviruses. 2013 Aug;29(8):1151-60. doi: 10.1089/AID.2012.0254. Epub 2013 May 6. PMID 23574474
- [Result] Yarasheski KE, Cade WT, Overton ET, Mondy KE, Hubert S, Laciny E, Bopp C, Lassa-Claxton S, Reeds DN. Exercise training augments the peripheral insulin-sensitizing effects of pioglitazone in HIV-infected adults with insulin resistance and central adiposity. Am J Physiol Endocrinol Metab. 2011 Jan;300(1):E243-51. doi: 10.1152/ajpendo.00468.2010. Epub 2010 Oct 19. PMID 20959530

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty four participants were enrolled from the AIDS Clinical Trials Unit and Infectious Diseases Clinics at Washington University School of Medicine in St. Louis, Missouri, USA. This was a prospective, two-group, random assignment study.
Pre-assignment Details: Exclusion criteria: medications or dietary supplements that affect metabolism (β-blocker, β-agonist, Ca2+ channel blocker, corticosteroid), neuromuscular disorder that affects metabolism or ability to exercise, consumed >3 alcohol drinks/wk, active Hep C or B, recreational-anabolic -appetite stimulant drugs, regular physical exercise.
Period: Overall Study
Arm/Group | Pioglitazone | Exercise Training
Started | 12 | 12
Completed | 12 | 8
Not Completed | 0 | 4
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | Exercise Training | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 42 (7) | 41 (6) | 42 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 9 | 12 | 21
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Myocardial Glucose Utilization Rate
Description: Radio-tracer (11C-glucose) and positron emission tomography quantification of myocardial glucose utilization rate. The rate at which glucose exits the blood, enters the muscle cells in the left ventricle, and is metabolized (ATP generation, glycolysis, glycogenolysis, or lactate production). Total glucose utilization rate in the left ventricle of the heart.
Time Frame: Weeks 0 and 16
Measure: Mean (Standard Error); unit: (nmol glucose/g heart muscle/min
Arm/Group | Pioglitazone | Exercise Training
Number analyzed (Participants) | 12 | 8
(nmol glucose/g heart muscle/min
  Week 0 | 109.6 (70.5) | 106.7 (69.0)
  Week 16 | 109.1 (55.2) | 87.2 (97.4)

2. Secondary Outcome: Myocardial Contractile Function During Diastole
Description: Echocardiographic quantification of (E/A) early to late diastolic filling velocity. Aria transfer blood to the ventricles in 2 steps:
  1. blood collected in the atria falls into the ventricles when the atrioventricular valves opens. In the left heart, the velocity at which the blood moves during this initial action is called the early or "E" filling velocity.
  2. residual blood in the atria, is emptied during diastole by atrial contraction. The velocity of the blood during atrial contraction is the "A" (for atrial) filling velocity. These are expressed as a ratio (E/A). If A exceeds E velocity (ratio <1.0) this is a clinical marker of diastolic dysfunction. This can occur when the left ventricular wall becomes so stiff as to impair proper filling, which can lead to diastolic heart failure.
Time Frame: Weeks 0 and 16
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Pioglitazone | Exercise Training
Number analyzed (Participants) | 12 | 8
ratio
  Week 0 | 1.4 (0.6) | 1.4 (0.3)
  Week 16 | 1.4 (0.5) | 1.5 (0.2)

3. Secondary Outcome: Myocardial Contractile Function During Systole
Description: Echocardiographic quantification of E' wall velocity during systole averaged at the lateral wall and septum
Time Frame: Weeks 0 and 16
Measure: Mean (Standard Error); unit: cm/sec
Arm/Group | Pioglitazone | Exercise Training
Number analyzed (Participants) | 12 | 8
cm/sec
  Week 0 | 12.7 (1.8) | 13.1 (2.4)
  Week 16 | 12.8 (1.6) | 13.6 (0.4)

4. Primary Outcome: Myocardial Glucose Utilization Rate Per Unit Insulin
Description: Radio-tracer (11C-glucose) and positron emission tomography quantification of myocardial glucose utilization rate per unit of plasma insulin. Total glucose utilization rate in the left ventricle of the heart expressed per unit of the circulating plasma insulin concentration.
Time Frame: Weeks 0 and 16
Measure: Mean (Standard Error); unit: (nmol glucose/g heart muscle/min/µU insu
Arm/Group | Pioglitazone | Exercise Training
Number analyzed (Participants) | 12 | 8
(nmol glucose/g heart muscle/min/µU insu
  Week 0 | 14.9 (22.1) | 11.9 (11.0)
  Week 16 | 15.7 (12.4) | 21.7 (40.8)

5. Primary Outcome: Myocardial Fatty Acid Utilization Rate
Description: Radio-tracer (11C-palmitate) and positron emission tomography quantification of myocardial fatty acid utilization rate. The rate at which palmitate exits the blood, enters the muscle cells in the left ventricle, and is metabolized (oxidation, re-esterification).
Time Frame: Weeks 0 and 16
Measure: Mean (Standard Error); unit: (nmol palmitate/g heart muscle/min
Arm/Group | Pioglitazone | Exercise Training
Number analyzed (Participants) | 12 | 8
(nmol palmitate/g heart muscle/min
  Week 0 | 119.3 (39.8) | 119.8 (48.7)
  Week 16 | 129.3 (34.5) | 130.4 (55.2)

6. Primary Outcome: Myocardial Fatty Acid Oxidation Rate
Description: Radio-tracer (11C-palmitate) and positron emission tomography quantification of myocardial fatty acid oxidation rate.
Time Frame: Weeks 0 and 16
Measure: Mean (Standard Error); unit: (nmol palmitate/g heart muscle/min
Arm/Group | Pioglitazone | Exercise Training
Number analyzed (Participants) | 12 | 8
(nmol palmitate/g heart muscle/min
  Week 0 | 92.4 (27.5) | 106.3 (49.6)
  Week 16 | 110.1 (31.7) | 97.5 (36.6)

7. Primary Outcome: Myocardial Fatty Acid Esterification
Description: Radio-tracer (11C-palmitate) and positron emission tomography quantification of myocardial fatty acid esterification as a % of total fatty acid extraction
Time Frame: Weeks 0 and 16
Measure: Mean (Standard Error); unit: (% of total fatty acid extraction)
Arm/Group | Pioglitazone | Exercise Training
Number analyzed (Participants) | 12 | 8
(% of total fatty acid extraction)
  Week 0 | 7 (7) | 4 (3)
  Week 16 | 4 (5) | 7 (5)

8. Secondary Outcome: Fasting Lipids and Lipoproteins
Description: fasting serum triglycerides, LDL-, and HDL-cholesterol concentrations
Time Frame: Week 0 and 16
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone | Exercise Training
Number analyzed (Participants) | 12 | 8
mg/dL
  triglycerides wk 0 | 199 (119) | 185 (58)
  triglycerides wk 16 | 182 (91) | 159 (33)
  LDL-cholesterol wk 0 | 115 (36) | 112 (26)
  LDL-cholesterol wk 16 | 97 (17) | 90 (24)
  HDL-cholesterol wk 0 | 38.9 (11.0) | 38.1 (8.4)
  HDL-cholesterol wk 16 | 38.8 (12.4) | 39.8 (21.8)

9. Secondary Outcome: Fasting Glucose Insulin and HOMA
Description: fasting plasma glucose, insulin concentrations and HOMA-insulin resistance
Time Frame: Week 0 and 16
Measure: Mean (Standard Error); unit: mg/dL µU/mL
Arm/Group | Pioglitazone | Exercise Training
Number analyzed (Participants) | 12 | 8
mg/dL µU/mL
  glucose (mg/dL) wk 0 | 102 (15) | 91.9 (9.5)
  glucose wk 16 | 95.3 (13) | 86.8 (8.2)
  insulin (µU/mL) wk 0 | 20.5 (25.7) | 14.8 (8.4)
  insulin wk 16 | 11.4 (9.6) | 11.8 (7.6)
  HOMA-IR wk 0 | 6.1 (10.4) | 3.3 (1.7)
  HOMA-IR wk 16 | 2.8 (2.7) | 2.6 (1.6)

ADVERSE EVENTS:
Arm/Group | Pioglitazone | Exercise Training
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/8
Other Adverse Events (participants affected / at risk) | 0/12 | 0/8

LIMITATIONS AND CAVEATS:
We did not perform the myocardial metabolic measurements under insulin-stimulated conditions (i.e. hyperinsulinemic clamps). Small number of participants and high measurement variability, efficacy was not found. Study ended to minimize risk/benefit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No